CLINICAL TRIAL: NCT03650881
Title: The Comparative Efficacy of an Over the Counter Light Therapy Mask vs Over the Counter Topical Benzoyl Peroxide 2.5% and Used in Combination With Over the Counter Adapalene Gel 0.1% for Mild to Moderate Acne
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible subjects were enrolled
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01725
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutrogena ® Light Therapy Acne Mask (MASK) (Experimental): Over-the-counter powered light-based device for the treatment of acne
  Interventions: Drug: Neutrogena ® Light Therapy Acne Mask (MASK)
- Topical benzoyl peroxide 2.5% gel and OTC adapalene (Active Comparator): Over-the-counter medication for the treatment of acne + 0.1% Adepalene Gel
  Interventions: Drug: Topical OTC benzoyl peroxide 2.5% gel and OTC adapalene

INTERVENTIONS:
Drug: Neutrogena ® Light Therapy Acne Mask (MASK) — Daily use of the OTC Neutrogena Light Therapy Acne Mask once daily for 10 minutes
  Arms: Neutrogena ® Light Therapy Acne Mask (MASK)
Drug: Topical OTC benzoyl peroxide 2.5% gel and OTC adapalene — Daily treatment with Reference Therapy OTC topical generic benzoyl peroxide 2.5% gel in the morning and OTC generic adapalene 0.1% gel at night
  Arms: Topical benzoyl peroxide 2.5% gel and OTC adapalene

SUMMARY:
This is a single-center prospective study of two standard-of-care treatments to evaluate the efficacy of the Neutrogena® Light Therapy Acne Mask an Over the Counter (OTC) Blue/Red light LED mask, as compared to the combination of topical OTC benzoyl peroxide 2.5% gel and OTC adapalene 0.1% gel, for the treatment of mild-to-moderate facial acne. This will be an investigator-blinded, randomized, 12-week study to observe these over the counter treatments. The two arms will be: (1) Neutrogena® Light Therapy Acne Mask (MASK), (2) topical OTC benzoyl peroxide 2.5% gel and OTC adapalene 0.1% gel (TOP). Both treatment groups in this study will also receive and use standardized, non-medicated cleansing and moisturizing products. All products will be purchased through commercial sources.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acne vulgaris as determined by the study physician
* Mild-to-moderate acne defined as a grade 2 or 3 on the FDA Investigator Global Acne Assessment (IGA) for Acne vulgaris (Appendix 1)19
* If female,

  * Negative urine pregnancy test at the time of enrollment and negative urine pregnancy tests at follow up visits
  * Agreement to comply with medically acceptable forms of birth control with heterosexual intercourse
* Agreement to comply with the study protocol and attend all study visits

Exclusion Criteria:

* Is unwilling to participate in the survey
* Outside of specified age range
* Patients with clear, almost clear acne, or severe acne defined as grade 0-1 or 4 on the IGA Scale
* Females who are pregnant or breastfeeding
* Known allergy to any ingredients in the test products or history of photosensitivity
* Pre-existing facial dermatologic conditions including excoriations that could interfere with the outcome of this study and quantification of acne lesions
* Excessive facial hair or scarring that could interfere with quantification of acne lesions
* Does not have decision making capacity

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
change in the Investigator Global Assessment (IGA) | 12 Weeks
  5 point assessment tool used to measure inflammation caused by acne

SECONDARY OUTCOMES:
change in Acne Q4 quality of life index score | 12 Weeks
  The Acne-QoL contains 19 questions organized into four domains (self-perception, role-social, roleemotional, and acne symptoms) which refer to facial acne. For all domains, higher scores reflect better HRQoL. The total score varies from zero to 114, distributed as follows: 0- 30 (self-perception), 0-24 (role-social), 0-30 (role-emotional), and 0-30 (acne symptoms).